CLINICAL TRIAL: NCT06870669
Title: The Effect of Progressive Relaxation Exercises Applied to First Year Nursing Students Before Clinical Practice on Perceived Stress, Psychological Resilience and Meaning of Life
Brief Title: The Effect of Progressive Relaxation Exercises by Nursing Students Before Clinical Practice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCBU-K-CEVIK-004
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Stress; Exercise
Keywords: Progressive Relaxation Exercises; Nursing; Students
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: progressive relaxation exercise

INTERVENTIONS:
Behavioral: progressive relaxation exercise — We will use progressive relaxation exercises to investigate the potential effects on first year nursing students' whose in the preclinical period of education.
  Arms: Intervention

SUMMARY:
Aim: We conducted this randomized controlled study to determine the effect of Progressive Relaxation Exercises practiced by first year nursing students before clinical practice on their perceptions of stress, psychological resilience and meaning of life.

Background: Progressive Relaxation Exercises has a positive effect on the person's mental/general health, life satisfaction and psychological well-being and enables the person to cope with stress.

Design: In this experimental randomized and controlled study including a control group, we administered a pre-test, post-test one and post-test two to the participating students.

Methods: We are planning the study with 40 first year nursing students in the intervention group, and 40 first year nursing students in the control group. The students in the intervention group took part in eight sessions of Progressive Relaxation Exercises for four weeks, twice a week. We used the Student Introduction Form, Perceived Stress Scale, Brief Psychological Resilience Scale and Meaning and Purpose of Life Scale to collect the study data.

ELIGIBILITY:
Inclusion Criteria:

Who did not have any diagnosed psychiatric diseases, Who had not done Progressive Relaxation Exercises and / or did not have any clinical experience previously were included

Exclusion Criteria:

Who withdrew from the study at any stage, Those who did not participate in the exercise sessions regularly Those who used another relaxation method during this period, Those who took antidepressants, Those who were unwilling to participate in the study, Those who lost one of their loved ones in the last 6 months were excluded from the research.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-03-13 (Estimated); Study Completion 2025-03-27 (Estimated)

PRIMARY OUTCOMES:
Stress | four weeks
  Stress of students was assessed with Perceived Stress Scale. Responses given to the items are rated on a 5-point Likert-type scale ranging from 0 to 4 (0- Never, 1-Almost Never, 2-Sometimes, 3-Quite often, 4-Very Often). Items 4, 5, 7 and 8 containing positive statements are reverse scored. The minimum and maximum scores that can be obtained from the PSS are 0 and 40, respectively. The higher the score is the higher the level of stress is.
psychological resilience | four weeks
  It is a 5-point Likert-type, 6-item, self-report measurement tool. After the reverse coded items in the scale are translated, high scores indicate high psychological resilience.
Meaning and Purpose of Life | four weeks
  Meaning of life of students was assessed with 17 items Meaning and Purpose of Life Scale. The options for the positive statements are scored as follows: strongly agree (5), agree (4), undecided (3), disagree (2), and strongly disagree (1). The negative statements are reverse scored. The options for the negative statements are scored as follows: strongly agree (1), agree (2), undecided (3), disagree (4) and strongly disagree (5).While the lowest possible score that can be obtained from the scale is 17, the highest possible score is 85. A high score indicates that the person's perception of the meaning and purpose of life is more positive whereas a low score indicates the person's perception of the meaning and purpose of life is more negative

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Yunusemre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No